CLINICAL TRIAL: NCT03391206
Title: Relationship Between Bioelectrical Impedance Utilization and Dietary Intake in the Analysis of Risk of Lymphedema in Breast Cancer Survivors: A Prospective Cross Sectional Study
Brief Title: Bioelectrical Impedance Utilization and Dietary Intake Relation in the Breast Cancer Related Lymphedema
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyung Seok Park, Clinical Assistant Professor, Severance Hospital
Other Study IDs: 4-2016-0149
Record Dates: First submitted 2017-10-11; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer Lymphedemas
Keywords: Breast cancer related lymphedemas; Sentinel Lymph Node Biopsy; Axillary Lymph Node Dissection; Bioelectrical Impedance Analysis; Dietary Fat
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- presence of BCRL: presence of breast cancer related lymphedema after surgical treatment using Inbody 720 and arm circumference measurement
  Interventions: Diagnostic Test: Inbody 720
- absence of BCRL: absence of breast cancer related lymphedema after surgical treatment using Inbody 720 and arm circumference measurement
  Interventions: Diagnostic Test: Inbody 720

INTERVENTIONS:
Diagnostic Test: Inbody 720 — We investigated the diagnostic accuracy of breast cancer related lymphedema diagnosed by bioimpedance analysis (Inbody 720) and arm circumference measurement..
  Other Names: bioelectrical impedance analysis

SUMMARY:
The purpose of this study was to investigate the clinical role of bioelectrical impedance analysis (BIA) and the relationship between the occurrence of breast cancer related lymphedema (BCRL) and dietary factors in breast cancer survivors who underwent surgical treatments.

DETAILED DESCRIPTION:
Breast cancer survivors are at risk of complications of breast cancer-related lymphedema (BCRL) after surgical treatments, which may negatively effect on the quality of life of breast cancer survivors. Lymphedema has been clinically diagnosed by determining that a limb is in fact swollen, and has arbitrarily been diagnosed in other etiologies. Limb circumference differences of 2 cm, a 200 mL or more in limb, or a 5% volume change are some of the objective ways that clinicians use to diagnose lymphedema. Although the arm circumference measurement method is a simple and frequently used clinical method, there is a disadvantage that the standardized reference point does not exist, the extracellular space can not be measured, and the sensitivity is also low. The lack of evidence-based diagnostic criteria to define lymphedema has presented tremendous difficulty in diagnosing lymphedema. It is important to define such criteria for early detection and treatment of lymphedema. Because of these limitations, many researchers are studying various methods for diagnosing lymphadenopathy and methods of bioelectrical impedance have been studied, recently.

Bioelectrical Impedance predicts body composition using the difference of electric conductivity by flowing a minute current to human body.This principle is used to diagnose the occurrence of lymphatic edema. In several studies, the single-frequency bioimpedance analysis (SFBIA) of the two arms obtained from bioelectrical impedance measurements was expressed as the ratio of the values of the operated and non-operated arms. However, it has not yet been clarified as a diagnostic method. Therefore, more studies are needed to establish a diagnosis method and a prediction method of lymphatic edema.

Various risk factors of lymphedema such as axillary lymph node dissection (ALND) and obesity have been studied for early prevention. However, there are no studies on the relationship between breast cancer related lymphedema, and dietary factors in breast cancer patients. The purpose of this study was to compare the diagnosis of lymphedema with the measurement of the arm circumference and the diagnosis of lymphedema through bioelectrical impedance values in order to clarify the clinical role of bioelectrical impedance method as a diagnostic method of lymphedema. To investigate the relationship between dietary factors, which are considered to be related to the occurrence of lymphedema, the investigators examined the frequency of dietary intake and analyzed the relationship between dietary factors and lymphatic edema.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients
* 20 years of age or older who survive after surgery and follow-up

Exclusion Criteria:

* Patients with bilateral breast cancer
* Male breast cancer patient
* Patients with a history of previous axillary surgery or radiation
* Recurrent breast cancer subjects
* Those who can not read or understand the written consent of an illiterate or foreigner
* Subjects who did not voluntarily decide to participate in this study or who did not sign a consent form
* The subjects who were judged inappropriate by the researcher to participate in this study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was conducted on women who were followed up at Severance Hospital for breast cancer survivors aged 20 years or older. Unilateral breast cancer patients at least 6 months after surgery were selected. They were voluntarily participated. The total number of patients recruited in this study was 250. Of these, 228 patients were enrolled, except for 10 patients with bilateral breast cancer, 10 patients with poor medical records, and 2 patients who did not measure bioelectrical impedance. 228 patients diagnosed lymphedema by arm circumference measurement.
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Brest cancer related lymphedema | At least six months after the surgical treatment
  Assessed by measuring the circumference at 15.0 centimeter below the acromion process in both arm and circumference difference of greater than or equal to 2.0 centimeter.

SECONDARY OUTCOMES:
BIA | At least six months after the surgical treatment
  bioelectrical impedance values
SFBIA ratio | At least six months after the surgical treatment
  single frequency bioelectrical impedance analysis
BMI | At least six months after the surgical treatment
  body mass index; weight in kilograms(kg) and height in meter(m) will be combined to report BMI in kg/m^2
WHR | At least six months after the surgical treatment
  waist-hip ratio; waist circumference in centimeter(cm) and hip circumference in centimeter(cm) will be combined to report WHR in cm/cm
Percent body fat | At least six months after the surgical treatment
  body fat mass in kilograms(kg) and weight in kilograms(kg) will be combined to report Percent body fat in kg/kg*100 (%)
Nutrient intake analysis | At least six months after the surgical treatment
  nutrient intake was analyzed by a nutrition analysis program (Can-Pro 5.0) through food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Seok Park, MD, Study Chair — Yonsei University College of Medicine, Korea
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim SM, Han Y, Kim SI, Park HS. Utilization of bioelectrical impedance analysis for detection of lymphedema in breast Cancer survivors: a prospective cross sectional study. BMC Cancer. 2019 Jul 8;19(1):669. doi: 10.1186/s12885-019-5840-9. PMID 31286884